CLINICAL TRIAL: NCT00096161
Title: Pentostatin and Donor Lymphocyte Infusion for Low Donor T-cell Chimerism After Hematopoietic Cell Transplantation - A Multi-center Trial
Brief Title: Pentostatin and Lymphocyte Infusion in Preventing Graft Rejection in Patients Who Have Undergone Donor Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Brenda Sandmaier, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1825.00; NCI-2010-00230 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1825.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P01CA078902 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Results first posted 2017-05-04 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Chronic Lymphocytic Leukemia; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Graft Versus Host Disease; Hodgkin Lymphoma; Myelodysplastic/Myeloproliferative Neoplasm; Non-Hodgkin Lymphoma; Plasma Cell Myeloma; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Graft vs Host Disease; Hodgkin Disease; Myelodysplastic-Myeloproliferative Diseases; Lymphoma, Non-Hodgkin; Multiple Myeloma; Waldenstrom Macroglobulinemia | interventions — Cyclosporine; Cyclosporins; Mycophenolic Acid; Pentostatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- pentostatin, DLI, mycophenolate mofetil, cyclosporine (Experimental): Group I (pentostatin, DLI): Patients receive pentostatin IV over 20-30 minutes on day -2 and DLI over 15-30 minutes on day 0. Treatment may repeat once beginning with an escalated or same CD3-dose at least 4 weeks if persistent donor T-cells are documented, no GvHD has developed, and the chimerism status worsens or, if chimerism status is unchanged after at least 8 weeks with two subsequent tests of chimerism 4 weeks apart.
  Group II (pentostatin, DLI, mycophenolate mofetil, cyclosporine): Patients receive treatment as in group I. Patients also receive cyclosporine PO BID on days -3 to 56 and mycophenolate mofetil PO QD on days 0 to 27. Treatment continues in the absence of GvHD.
  Interventions: Drug: Cyclosporine; Drug: Mycophenolate Mofetil; Drug: Pentostatin; Biological: Therapeutic Allogeneic Lymphocytes

INTERVENTIONS:
Drug: Cyclosporine — Given PO
  Other Names: 27-400; Ciclosporin; CsA; Cyclosporin; Cyclosporin A; Neoral; OL 27-400; Sandimmun; Sandimmune; SangCya
Drug: Mycophenolate Mofetil — Given PO
  Other Names: Cellcept; MMF
Drug: Pentostatin — Given IV
  Other Names: (R)-3-(2-Deoxy-.beta.-D-erythro-pentofuranosyl)-3,6,7, 8-tetrahydroimidazo[4,5-d][1,3]diazepin-8-ol; 2'-Deoxycoformycin; CI-825; Co-Vidarabine; Covidarabine; DCF; Deoxycoformycin; Nipent; PD-81565; Pentostatine
Biological: Therapeutic Allogeneic Lymphocytes — Given IV
  Other Names: Allogeneic Lymphocytes

SUMMARY:
This phase II trial studies pentostatin and donor lymphocyte infusion in preventing graft rejection in patients who have undergone donor stem cell transplant. Giving pentostatin and an infusion of the donor's T cells (donor lymphocyte infusion) after a donor stem cell transplant may stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving pentostatin before donor lymphocyte infusion may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and efficacy of the combined use of pentostatin and donor lymphocyte infusion (DLI) in patients with low or falling donor T-cell chimerism to prevent graft rejection after transplantation both from matched related donors (MRDs) or unrelated donors (URDs).

SECONDARY OBJECTIVES:

I. To determine the incidence of graft-versus-host disease (GvHD) infections and disease response, if persistent disease is present.

OUTLINE: This is a dose-escalation study of donor lymphocyte infusion.

GROUP I: Patients receive pentostatin intravenously (IV) over 20-30 minutes on day -2 and DLI over 15-30 minutes on day 0. Treatment may repeat once beginning with an escalated or same cluster of differentiation (CD)3-dose at least 4 weeks if persistent donor T-cells are documented, no GvHD has developed, and the chimerism status worsens or, if chimerism status is unchanged after at least 8 weeks with two subsequent tests of chimerism 4 weeks apart.

GROUP II (initiated if patients in group I do not achieve sustained engraftment and improved chimerism): Patients receive treatment as in group I. Patients also receive cyclosporine orally (PO) twice daily (BID) on days -3 to 56 and mycophenolate mofetil PO once daily (QD) on days 0 to 27. Treatment continues in the absence of GvHD.

After completion of study treatment, patients are followed up every 6 months for 2 years and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients having received a preceding allogeneic transplantation from either a human leukocyte antigen (HLA)-matched related or unrelated donor are eligible for this protocol

  * Related donor: HLA genotypically identical at least at one haplotype and may be phenotypically or genotypically identical at the allele level at HLA A, B, C, DRB1, and DQB1
  * Unrelated donor who are prospectively:

    * Matched for HLA-A, B, C, DRB1 and DQB1 by high resolution typing; OR
    * Only a single allele disparity will be allowed for HLA-A, B, or C as defined by high resolution typing
* Patients with less than 50% donor CD3 peripheral blood chimerism on two separate, consecutive evaluations; the two evaluations must be at least 14 days apart OR patients with absolute decreases of donor CD3 peripheral blood chimerism of >= 20% if the second test shows < 50% donor CD3 cells; the two evaluations must be at least 14 days apart
* Patients with evidence of disease are only eligible if the disease is stable (or persistent) in comparison to the status prior to transplantation
* Patients must be tapered off systemic steroids to a dosage of less than or equal to 0.25 mg/kg/day
* Patients must have persistent donor CD3 cells (>= 5% donor CD3 cells by a deoxyribonucleic acid [DNA]-based assay that compares the profile of amplified fragment length polymorphisms [ampFLP] [or fluorescent in situ hybridization (FISH) studies or variable number of tandem repeats (VNTR)])
* DONOR: Alternatively to a fresh unmodified leukapheresis product, previously collected cryopreserved peripheral blood stem cells (PBSC) after mobilization with G-CSF or cryopreserved unmodified leukapheresis product from the original donor can be used; if cryopreserved product is not available, the following criteria apply for the DLI product:
* DONOR: Original donor of hematopoietic cell transplantation
* DONOR: Donor must give consent to leukapheresis
* DONOR: Donor must have adequate veins for leukapheresis or agree to placement of central venous catheter (femoral or subclavian)
* DONOR: Donor must be medically fit to undergo the apheresis procedure (institutional guidelines for apheresis)

Exclusion Criteria:

* Current grade II to IV acute GVHD or extensive chronic GVHD
* Karnofsky score < 50%

  * Pediatric criteria

    * Lansky play-performance score < 40
* Evidence of relapse or progression of disease after transplantation
* Prior recipient of cord blood
* DONOR: Donors who are not suitable for medical reasons to donate peripheral blood mononuclear cells (PBMC) by continuous centrifugation according to the criteria of the American Association of Blood Banks (AABB)
* DONOR: Pregnancy
* DONOR: Human immunodeficiency virus (HIV) or human T-lymphotrophic virus (HTLV) infection
* DONOR: Recent immunization may require a delay

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2003-05 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Sandmaier, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (5):
- United States (4):
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - VA Puget Sound Health Care System, Seattle, Washington
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
- University of Torino, Torino, Italy

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1A (Pentostatin, DLI Dose Level 1): Patients receive pentostatin IV over 20-30 minutes on day -2 and DLI (1x10^7 CD3+ cells/kg) over 15-30 minutes on day 0. Treatment may repeat once beginning with an escalated or same CD3-dose at least 4 weeks if persistent donor T-cells are documented, no GvHD has developed, and the chimerism status worsens or, if chimerism status is unchanged after at least 8 weeks with two subsequent tests of chimerism 4 weeks apart.
  Pentostatin: Given IV
  Therapeutic Allogeneic Lymphocytes: Given IV
- Group 1B (Pentostatin, DLI Dose Level 2): Patients receive pentostatin IV over 20-30 minutes on day -2 and DLI (3x10^7 CD3+ cells/kg) over 15-30 minutes on day 0. Treatment may repeat once beginning with an escalated or same CD3-dose at least 4 weeks if persistent donor T-cells are documented, no GvHD has developed, and the chimerism status worsens or, if chimerism status is unchanged after at least 8 weeks with two subsequent tests of chimerism 4 weeks apart.
  Pentostatin: Given IV
  Therapeutic Allogeneic Lymphocytes: Given IV
- Group 2C (Pentostatin, DLI Dose Level 1, Add'l IS): Patients receive treatment as in group 1A. Patients also receive cyclosporine PO BID on days -3 to 56 and mycophenolate mofetil PO QD on days 0 to 27. Treatment continues in the absence of GvHD.
  Pentostatin: Given IV
  Therapeutic Allogeneic Lymphocytes: Given IV
- Group 2D (Pentostatin, DLI Dose Level 2, Add'l IS): Patients receive treatment as in group 1B. Patients also receive cyclosporine PO BID on days -3 to 56 and mycophenolate mofetil PO QD on days 0 to 27. Treatment continues in the absence of GvHD.
  Pentostatin: Given IV
  Therapeutic Allogeneic Lymphocytes: Given IV
Period: Overall Study
Arm/Group | Group 1A (Pentostatin, DLI Dose Level 1) | Group 1B (Pentostatin, DLI Dose Level 2) | Group 2C (Pentostatin, DLI Dose Level 1, Add'l IS) | Group 2D (Pentostatin, DLI Dose Level 2, Add'l IS)
Started | 20 | 10 | 6 | 0
Completed | 20 | 10 | 6 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No subjects were enrolled onto Group 2D because the dose escalation was not triggered before the study closed to accrual.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1A (Pentostatin, DLI Dose Level 1) | Group 1B (Pentostatin, DLI Dose Level 2) | Group 2C (Pentostatin, DLI Dose Level 1, Add'l IS) | Group 2D (Pentostatin, DLI Dose Level 2, Add'l IS) | Total
Number analyzed (Participants) | 20 | 10 | 6 | 0 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 7 | 4 | 0 | 28
  >=65 years | 3 | 3 | 2 | 0 | 8
Age, Continuous [Median (Full Range); unit: years] | 55 [44 to 67] | 59.3 [35 to 72] | 60.3 [47 to 69] |  | 56.9 [35 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 |  | 5
  Male | 18 | 8 | 5 |  | 31
Region of Enrollment [Number; unit: participants]
  United States | 20 | 10 | 6 |  | 36

OUTCOME MEASURES:

1. Primary Outcome: Percentage Patients With an Increase of at Least 10 Percentage Points in Donor T-cell Chimerism
Description: A regimen will be considered successful if 20 patients are enrolled, at least 13 demonstrate improved chimerism. If fewer than 5 patients have shown improvement in chimerism then it can be at least 75% confident that the true rate of improvement is less than 0.53. Enrollment to the regimen will stop and the next regimen will be opened. Enrollment to a regimen may also be stopped at any time it becomes impossible to achieve 5 of 10 or 13 of 20 successful improvements.
  "Chimerism" in hematopoietic cell transplant derives from this idea of a "mixed" entity, referring to someone who has received a transplant of genetically different tissue. A test for chimerism after a hematopoietic cell transplant involves identifying the genetic profiles of the recipient and of the donor and then evaluating the extent of mixture in the recipient's blood cells or marrow cells.
Time Frame: From the time of enrollment maintained to day 56 after the last DLI, up to Day 112
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Group 1A (Pentostatin, DLI Dose Level 1) | Group 1B (Pentostatin, DLI Dose Level 2) | Group 2C (Pentostatin, DLI Dose Level 1, Add'l IS) | Group 2D (Pentostatin, DLI Dose Level 2, Add'l IS)
Number analyzed (Participants) | 20 | 10 | 6 | 0
percentage of participants | 60 | 30 | 33.3 |

2. Primary Outcome: Incidence of Grade IV Acute GVHD
Description: Clinical Stage of acute GVHD according to Organ System
  Skin:
  1. - Maculopapular rash <25% of body surface
  2. - Maculopapular rash 25-50% of body surface
  3. - Maculopapular rash >50% body surface area or generalized erythroderma
  4. - Generalized erythroderma with bullous formation and desquamation
  Liver:
  1. - Bilirubin 2-3 mg/dl
  2. - Bilirubin 3.1-6 mg/dl
  3. - Bilirubin 6.1-15 mg/dl
  4. - Bilirubin >15 mg/dl
  Gut:
  1. - >500-1000 mL diarrhea per day or (nausea, anorexia or vomiting with biopsy (EGD) confirmation of upper GI GVHD
  2. - >1000 -1500 mL diarrhea per day
  3. - >1500 mL diarrhea per day
  4. - >1500 mL diarrhea per day plus severe abdominal pain with or without ileus
  Overall Clinical Grading of Severity of acute GVHD Grade IV: 0-4 Skin, 2-4 Liver, and/or 2-4 GI
Time Frame: Within 100 days after the last DLI
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Group 1A (Pentostatin, DLI Dose Level 1) | Group 1B (Pentostatin, DLI Dose Level 2) | Group 2C (Pentostatin, DLI Dose Level 1, Add'l IS) | Group 2D (Pentostatin, DLI Dose Level 2, Add'l IS)
Number analyzed (Participants) | 20 | 10 | 6 | 0
percentage of participants | 5 | 0 | 0 |

3. Secondary Outcome: Incidence of GVHD
Description: Percentage patients with acute or chronic GVHD.
  The diagnosis of chronic GVHD requires at least one manifestation that is distinctive for chronic GVHD as opposed to acute GVHD. In all cases, infection and others causes must be ruled out in the differential diagnosis of chronic GVHD.
Time Frame: 1 year after DLI
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Group 1A (Pentostatin, DLI Dose Level 1) | Group 1B (Pentostatin, DLI Dose Level 2) | Group 2C (Pentostatin, DLI Dose Level 1, Add'l IS) | Group 2D (Pentostatin, DLI Dose Level 2, Add'l IS)
Number analyzed (Participants) | 20 | 10 | 6 | 0
percentage of participants
  aGVHD | 20 | 0 | 0 |
  cGVHD | 50 | 20 | 16.7 |

4. Secondary Outcome: Incidence of Infections
Time Frame: 100 days after DLI
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Group 1A (Pentostatin, DLI Dose Level 1) | Group 1B (Pentostatin, DLI Dose Level 2) | Group 2C (Pentostatin, DLI Dose Level 1, Add'l IS) | Group 2D (Pentostatin, DLI Dose Level 2, Add'l IS)
Number analyzed (Participants) | 20 | 10 | 6 | 0
percentage of participants | 80 | 70 | 33.3 |

5. Secondary Outcome: Incidence of Relapse/Progression
Description: CML Acquisition of a new cytogenetic abnormality and/or development of accelerated phase or blast crisis. Criteria for accelerated phase: unexplained fever >38.3° C, new clonal cytogenetic abnormalities in addition to a single Ph-positive chromosome, BM blasts and promyelocytes >20%.
  AML, ALL, CMML >30% BM blasts w/ deteriorating performance status, or worsening of anemia, neutropenia, or thrombocytopenia.
  CLL Progressive disease: ≥1 of: physical exam/imaging studies (nodes, liver, and/or spleen) ≥50% increase or new, circulating lymphocytes by morphology and/or flow cytometry ≥50% increase, and lymph node biopsy w/ Richter's transformation.
  NHL >25% increase in the sum of the products of the perpendicular diameters of marker lesions, or the appearance of new lesions.
  MM
  ≥100% increase of the serum myeloma protein from its lowest level, or reappearance of myeloma peaks that had disappeared w/ tx; or definite increase in the size/number of plasmacytomas or lytic bone lesions.
Time Frame: 1 year after DLI
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Group 1A (Pentostatin, DLI Dose Level 1) | Group 1B (Pentostatin, DLI Dose Level 2) | Group 2C (Pentostatin, DLI Dose Level 1, Add'l IS) | Group 2D (Pentostatin, DLI Dose Level 2, Add'l IS)
Number analyzed (Participants) | 20 | 10 | 6 | 0
percentage of participants | 45 | 20 | 33.3 |

6. Secondary Outcome: Survival
Description: Percentage patients surviving.
Time Frame: 1 year after DLI
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Group 1A (Pentostatin, DLI Dose Level 1) | Group 1B (Pentostatin, DLI Dose Level 2) | Group 2C (Pentostatin, DLI Dose Level 1, Add'l IS) | Group 2D (Pentostatin, DLI Dose Level 2, Add'l IS)
Number analyzed (Participants) | 20 | 10 | 6 | 0
percentage of participants | 60 | 90 | 66.7 |

ADVERSE EVENTS:
Time Frame: AEs: Conditioning through Day 100; SAEs: Conditioning through Day 200
Description: One incident of GVHD was incorrectly reported as an SAE, as it is an expected complication of DLI. This patient outcome is recorded under deaths.
Arm/Group | Group 1A (Pentostatin, DLI Dose Level 1) | Group 1B (Pentostatin, DLI Dose Level 2) | Group 2C (Pentostatin, DLI Dose Level 1, Add'l IS) | Group 2D (Pentostatin, DLI Dose Level 2, Add'l IS)
Serious Adverse Events (participants affected / at risk) | 6/20 | 0/10 | 0/6 | 0/0
Other Adverse Events (participants affected / at risk) | 10/20 | 2/10 | 2/6 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1A (Pentostatin, DLI Dose Level 1) (N=20) | Group 1B (Pentostatin, DLI Dose Level 2) (N=10) | Group 2C (Pentostatin, DLI Dose Level 1, Add'l IS) (N=6) | Group 2D (Pentostatin, DLI Dose Level 2, Add'l IS) (N=0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GVHD (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1A (Pentostatin, DLI Dose Level 1) (N=20) | Group 1B (Pentostatin, DLI Dose Level 2) (N=10) | Group 2C (Pentostatin, DLI Dose Level 1, Add'l IS) (N=6) | Group 2D (Pentostatin, DLI Dose Level 2, Add'l IS) (N=0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Cardiac troponin I increased (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Forced expiratory volume decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Ileal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other, (Pancytopenia) (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestine infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes